CLINICAL TRIAL: NCT04816266
Title: Comparative Study Between Pentacam and IOL Master in Measuring Anterior Chamber Depth
Brief Title: Comparative Study in Measuring Anterior Chamber Depth
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Engy Adel Fayez Demian, Principal investigator, Assiut University
Other Study IDs: Anterior chamber depth
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Error, Refractive
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Myopic patients
  Interventions: Device: Iol master; Device: Pentacam
- Hypermetropic patients
  Interventions: Device: Iol master; Device: Pentacam
- Emmetropic people
  Interventions: Device: Iol master; Device: Pentacam

INTERVENTIONS:
Device: Iol master — Iol master measures the distance between anterior pole of the cornea and the anterior surface of the lens to calculate the anterior chamber depth
Device: Pentacam — The Pentacam HR calculates Anterior chamber depth from the corneal endothelial layer along a line from the apex of the cornea to the anterior surface of the lens

SUMMARY:
Measuring parameters of anterior segment of the eye accurately is important for diagnosing variety of diseases and for cataract surgeries, glaucoma, refractive surgeries and post-operative follow-up. One of the anterior segment parameters is the anterior chamber depth.

The anterior chamber depth (ACD) measurement provides valuable information in different fields in ophthalmology. Firstly, it is important for the new theoretical biometric formulas used to calculate the power of intraocular lenses (IOLs) .Secondly, phakic IOL implantation requires precise ACD measurement for both surgical planning and IOL power calculation. Thirdly, the ACD is also implicated as a screening risk factor for glaucoma. Additionally, precise ACD measurement is thought to be important to the accurate determination of the optic zone ablation diameter for keratorefractive surgery, as well as for the analysis of postoperative ACD changes.

Different technologies are used in measurement of the anterior chamber depth Such as pentacam and iol maste

DETAILED DESCRIPTION:
IOL master :

Optical biometry by the IOL Master was introduced in the United Kingdom in 1999.Its technology is based on laser interfer-ometry with partial coherent light, termed as Partial Coherence Interferometry (PCI).The device uses the principle of PCI to measure the axial length of the eye.While uses a slit-beam photo-graphic technique for ACD measurements For keratometry measurement, six light spots are projected hexagonally on the cornea .The device records the reflection of these images measuring the separation of the opposite pairs of light spots and calculating the corneal radii and toroidal surface curvature. The mean of the taken measurements is considered the corneal power . The displayed K1 and K2 represent the average keratometry values at two major perpendicular meridians .For ACD measurement, the IOL Master directs a slit beam of light 0.7mm wide through the anterior segment at an angle of 38º to the visual axis.The internal software measures the distance between anterior pole of the cornea and the anterior surface of the lens to calculate the ACD . The device takes five ACD measurements in rapid succession; the mean of these readings are taken as the ACD value . For WTW measurement, a digital grey-scale photograph of the anterior surface of the eye is taken after focusing on the iris. The limbus is then detected automatically and the WTW distance is measured

Pentacam :

The Pentacam obtains images of the anterior segment by a rotating Scheimpflug blue Light Emitting Diode (LED) with a wavelength of 475nm. It acquires 50 images in a duration of approximately two seconds. It extracts about 2,760 true elevation points from the obtained images which in turn generates 1 38,000 true elevation points for the both front and back corneal surfacesand from limbus to limbus, including the central part of the cornea . There for, it calculates k-readings of the cornea. The Pentacam HR calculates ACD from the corneal endothelial layer along a line from the apex of the cornea to the anterior surface of the lens . Horizontal WTW was measured by manual placement of callipers on the Scheimpflug image of the horizontal plane of the examined eye; callipers are placed on the corneo-scleral junction then a line is automat-ically drawn between the two points . The length of this line represents the WTW value

ELIGIBILITY:
Inclusion Criteria:

* presenting for glasses
* asking for refractive surgery

Exclusion Criteria:

* severe corneal scarring or opacity
* patients with corneal dystrophy
* patients with keratoconus
* patients with previous ocular surgery
* patients with ocular trauma
* patients with uveitis

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: People between eighteen and forty years seeking for refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Comparison between values of anterior chamber depth obtained by different devices | One year
  Measuring Anterior chamber depth by Pentacam and iol master in eyes with different refractive errors